CLINICAL TRIAL: NCT02137187
Title: A Randomized Controlled Trial of Atrioventricular (AV) Junction Ablation and Biventricular Pacing Versus Optimal Pharmacological Therapy in Patients With Permanent Atrial Fibrillation
Brief Title: Atrioventricular Junction Ablation and Biventricular Pacing for Atrial Fibrillation and Heart Failure
Acronym: APAF-CRT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Prevenzione Malattie Cardiovascolari N. e V. Corbella (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPMCV-01-14
Record Dates: First submitted 2014-05-03; First posted 2014-05-13 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2020-07

CONDITIONS: Permanent Atrial Fibrillation
Keywords: Atrial fibrillation; Heart failure; Catheter ablation; Cardiac resynchronization therapy; Implantable defibrillator
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure | interventions — Cardiac Resynchronization Therapy; Defibrillators, Implantable

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug therapy (Experimental): Control Arm: optimized drug therapy (plus implantable defibrillator (ICD) according to guidelines)
  Interventions: Drug: Optimized drug therapy; Device: ICD
- Device: AV junction ablation & CRT (Active Comparator): AV junction ablation + CRT (CRT-P or CRT-D according to guidelines) + optimized drug therapy
  Interventions: Procedure: AV junction ablation; Device: CRT; Drug: Optimized drug therapy; Device: ICD

INTERVENTIONS:
Procedure: AV junction ablation — AV junction ablation
  Other Names: AV nodal ablation
  Arms: Device: AV junction ablation & CRT
Device: CRT — Implantation of device for pacing and cardiac resynchronization therapy (CRT-P or CRT-D according to guidelines)
  Other Names: Cardiac resynchronization therapy
  Arms: Device: AV junction ablation & CRT
Drug: Optimized drug therapy — Optimized drug therapy for heart failure and atrial fibrillation rate control
  Other Names: Pharmacological therapy
Device: ICD — Implantable defibrillator (in control Group or in association with CRT in study Group) according to guidelines
  Other Names: Implantable defibrillator

SUMMARY:
There is evidence of superiority of AV junction ablation strategy over pharmacological therapy only for symptoms of atrial fibrillation, but not for heart failure, hospitalization, morbidity and mortality. Hypothesis of trial is that AV junction ablation is superior to pharmacological therapy as regard hospitalization and mortality

DETAILED DESCRIPTION:
Prospective randomized, controlled, investigator-initiated trial which consists of two specific consecutive(overlapped) phases:

"Morbidity trial" (APAF-CRT morbidity). Small size (280 pts), follow-up 24 months. Primary endpoint: combined of mortality due to heartfailure, hospitalization for heart failure or atrial fibrillation or worsening heart failure. Predefined subgroup analysis for patients with ejection fraction ≤35% versus >35%

"Mortality trial" (APAF-CRT mortality). Large size (pts included in morbidity trial plus additional ~1500 pts, long-term follow-up (at least 4 years). Primary endpoint: total mortality. Predefined subgroup analysis for patients with ejection fraction ≤35% versus >35%

ELIGIBILITY:
Inclusion Criteria:

To be eligible, each patient must be in the following condition:

1. Permanent atrial fibrillation (>6 months) which has been considered unsuitable for ablation or failed ablation
2. Narrow QRS ≤ 110 ms
3. Severely symptomatic (atrial fibrillation-related symptoms), refractory to drug therapy for rate control
4. At least one hospitalization related to atrial fibrillation and/or heart failure in the previous year (see definition below)

Exclusion Criteria:

1. New York Heart Association (NYHA) class IV and systolic blood pressure <80 mmHg despite optimized therapy;
2. severe concomitant non-cardiac disease;
3. need for surgical intervention;
4. myocardial infarction within the previous 3 months;
5. previous implanted devices (PM/ICD/CRT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1830 (Estimated)
Dates: Start 2014-10-15 (Actual); Primary Completion 2021-05-15 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Combined end-point | Upto 3 years
  "Morbidity trial" end-points Primary end-point: a combined of (1) mortality due to heart failure, (2) hospitalization for heart failure or uncontrolled intolerable atrial fibrillation, or (3) worsening heart failure

SECONDARY OUTCOMES:
Major clinical events | Up to 3 years
  "Morbidity trial" end-points Secondary end-points: total mortality, total hospitalizations, hospitalization for heart failure and/or atrial fibrillation and worsening heart failure.
Major clinical events | Up to 5 years
  "Mortality trial" end-points Secondary end-point: cardiovascular mortality and hospitalization for heart failure or uncontrolled intolerable atrial fibrillation

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Marsano, MD, Study Director — Centro Prevenzione Malattie Cardiovascolari N. e V. Corbella
Locations (1):
- Department of Cardiology, Ospedali del Tigullio, Lavagna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chatterjee NA, Upadhyay GA, Ellenbogen KA, McAlister FA, Choudhry NK, Singh JP. Atrioventricular nodal ablation in atrial fibrillation: a meta-analysis and systematic review. Circ Arrhythm Electrophysiol. 2012 Feb;5(1):68-76. doi: 10.1161/CIRCEP.111.967810. Epub 2011 Dec 20. PMID 22187425
- [Result] Brignole M, Botto G, Mont L, Iacopino S, De Marchi G, Oddone D, Luzi M, Tolosana JM, Navazio A, Menozzi C. Cardiac resynchronization therapy in patients undergoing atrioventricular junction ablation for permanent atrial fibrillation: a randomized trial. Eur Heart J. 2011 Oct;32(19):2420-9. doi: 10.1093/eurheartj/ehr162. Epub 2011 May 23. PMID 21606084
- [Derived] Brignole M, Pentimalli F, Palmisano P, Landolina M, Quartieri F, Occhetta E, Calo L, Mascia G, Mont L, Vernooy K, van Dijk V, Allaart C, Fauchier L, Gasparini M, Parati G, Soranna D, Rienstra M, Van Gelder IC; APAF-CRT Trial Investigators. AV junction ablation and cardiac resynchronization for patients with permanent atrial fibrillation and narrow QRS: the APAF-CRT mortality trial. Eur Heart J. 2021 Dec 7;42(46):4731-4739. doi: 10.1093/eurheartj/ehab569. PMID 34453840
- [Derived] Brignole M, Pokushalov E, Pentimalli F, Palmisano P, Chieffo E, Occhetta E, Quartieri F, Calo L, Ungar A, Mont L; APAF-CRT Investigators. A randomized controlled trial of atrioventricular junction ablation and cardiac resynchronization therapy in patients with permanent atrial fibrillation and narrow QRS. Eur Heart J. 2018 Dec 1;39(45):3999-4008. doi: 10.1093/eurheartj/ehy555. PMID 30165479